CLINICAL TRIAL: NCT02222987
Title: Influence of Oral Doses of 75 mg Clopidogrel on the Pharmacodynamics and Safety of Oral Doses of 100 mg Terbogrel Bid Over 8 Days in Healthy Male Subjects. An Intra-individual, Open Trial.
Brief Title: Influence of Clopidogrel on the Pharmacodynamics and Safety of Terbogrel in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 528.23
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — terbogrel; Clopidogrel

ARMS (3):
- Terbogrel (Active Comparator)
  Interventions: Drug: Terbogrel
- Terbogrel with Clopidogrel (Experimental)
  Interventions: Drug: Terbogrel; Drug: Clopidogrel
- Clopidogrel (Active Comparator)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Terbogrel
  Arms: Terbogrel; Terbogrel with Clopidogrel
Drug: Clopidogrel
  Arms: Clopidogrel; Terbogrel with Clopidogrel

SUMMARY:
Study to assess the influence of 75 mg clopidogrel on the pharmacodynamics and safety of 100 mg terbogrel bid.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Healthy male subjects
* Age >= 18 and <= 45 years
* Broca >= -20% and <= +20 %

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of

  * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * any bleeding disorder including prolonged or habitual bleeding
  * other hematologic disease
  * cerebral bleeding (e.g. after car accident)
  * commotio cerebri
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months days prior to administration or during the trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol (> 60 g/day) abuse
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the reference range of clinical relevance
* History of any familial bleeding disorder
* Thrombocytes < 150000/µl

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 1999-02; Primary Completion 1999-03 (Actual)

PRIMARY OUTCOMES:
Change in inhibition of platelet aggregation in platelet rich plasma (PRP) | baseline, up to day 17
Change in thromboxane receptor occupancy (TRO) | baseline, up to day 17
Change in 6-keto-prostaglandinF-1-alpha | baseline, up to day 17
Change in thromboxan synthesis inhibition (TSI) | baseline, up to day 17

SECONDARY OUTCOMES:
Plasma levels of terbogrel | up to day 17
Number of patients with adverse events | up to day 17
Change in bleeding time | baseline, up to day 17
Change in systolic and diastolic blood pressure | baseline, up to day 17
Change in pulse rate | baseline, up to day 17
Number of patients with haematuria | up to day 17
  dipstick test
Number of patients with positive Haemoccult test | up to day 17
Number of patients with clinically significant laboratory findings | up to day 17